CLINICAL TRIAL: NCT04245124
Title: Validation of Cognitive Enhancement Techniques for Mild Traumatic Brain Injury
Acronym: VoCET-mTBI
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: The Defense and Veterans Brain Injury Center (U.S. Federal Agency)
Collaborators: The University of Texas at Dallas (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: NHCP.2020.0006
Record Dates: First submitted 2019-11-08; First posted 2020-01-28 (Actual); Last update posted 2021-02-03 (Actual); Status verified 2021-02

CONDITIONS: Mild Traumatic Brain Injury
Keywords: COGNITIVE REHABILITATION
MeSH Terms: conditions — Brain Concussion

STUDY DESIGN:
Intervention Model Description: Primary Aim: Difference in Cognitive and Neurophysiological Function between SMART and TCR. Multilevel mixed-effect modeling will be conducted for Aim 1 with treatment modality (SMART vs. TCR) as the independent variable. This approach will take into consideration between-subject variance based on randomized group, as well as within-subject variance for repeated measures. Primary analyses will be based on intention to treat, and we will leverage the statistical power of multilevel modeling to handle missing follow-up data. Outcome will be assessed as change in GDS over time. A significant p-value of 0.05 will be used to assess the main effects.
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- SMART INTERVENTION (Experimental): N= 81 20 HOURS THERAPY IMMEDIATE POST TREATMENT EVALUATION 3 MONTH POST TREATMENT EVALUATION
  Interventions: Other: Strategic Memory Advanced Reasoning Training
- TCR (Experimental): N= 81 60 HOURS THERAPY IMMEDIATE POST TREATMENT EVALUATION 3 MONTH POST TREATMENT EVALUATION
  Interventions: Other: Traditional Cognitive Rehabilitation

INTERVENTIONS:
Other: Strategic Memory Advanced Reasoning Training — SMART focuses on three metacognitive strategies: Strategic Attention, Integrated Reasoning and Innovation.
  Arms: SMART INTERVENTION
Other: Traditional Cognitive Rehabilitation — Participants randomized to the TCR condition will participate in a clinician-directed intervention that provides manualized, traditional clinician-directed cognitive rehabilitation that was developed for the SCORE trial (Cooper et al., 2017)
  Arms: TCR

SUMMARY:
With an average of 21,000 diagnosed brain injuries each year among military personnel, traumatic brain injury (TBI) remains a major health concern for the United States Military Health System. Mild traumatic brain injury (mTBI) is the most common type of brain injury sustained by military personnel and may result in chronic cognitive impairment.Unfortunately, many service members (SMs) have a history of multiple head injuries as well as psychological co-morbidities that negatively influence recovery. Advances in treatment options for cognitive rehabilitation following mTBI have been of increasing interest to the medical community and may increase treatment efficacy for injured SMs to ensure force readiness.

Cognitive Rehabilitation (CR) for severe brain injury focuses on compensatory strategies for activities of daily living such as using lists to remember grocery items or reminders to take medications and attend medical appointments. Research has shown CR interventions to have considerable effectiveness in the acute and sub-acute phase of recovery after severe TBI. But there is insufficient evidence that they improve rates of individuals returning to work, independence in activities of daily living (ADL), community re-integration, or quality of life.

DETAILED DESCRIPTION:
Cognitive Rehabilitation for mild brain injury has shown some modest evidence of effectiveness. CR interventions for mTBI typically focus on compensating for subjective and functional cognitive complaints. A number of recent studies have examined the use of compensatory CR approaches for individuals (primarily military veterans) diagnosed with mild cognitive impairment from a likely mTBI. These interventions taught individuals adaptive functional skills (e.g., cognitive mnemonics) and highlighted use of external aids such as smart phone scheduling/reminder applications. A randomized control trial that included 16 veterans with TBI (mixed mild and moderate severity), found this compensatory CR intervention was effective at reducing overall symptoms, but did not impact cognitive performance or work-outcomes. In a secondary study, there was some evidence that the compensatory CR intervention improved memory at 6 months post-treatment and quality of life at 12 months but there was not a consistent pattern of improvement compared to controls.

Generalizability from civilian and veteran communities to active duty SMs may pose some unique and unexplored factors as the goal of treatment is not remediation of common activities of daily living (e.g., remembering appointments) but in contrast, the goal is military readiness needed for worldwide deployability to potential wartime environments (e.g., "cognitive readiness").

ELIGIBILITY:
Inclusion Criteria:

* • Male or female ages 18 years or older

  * Active duty military personnel
  * History of mTBI: participants will have a history of at least one mTBI sustained >3 months previously based on criteria of the DoD diagnostic criteria (Department of Veterans Affairs and Department of Defense, 2016). This specifies an external force to the head which resulted in physiological dysfunction of the brain as manifested by one or more of the following acute symptoms:

    1. Any loss of consciousness (not to exceed 30 minutes)
    2. Any loss of memory for the events immediately before or after the injury (not to exceed 1 day)
    3. Any alteration of consciousness or change in mental state (not to exceed 24 hours)
  * Persistent Post-Concussive Symptoms: Participants will endorse elevated neurobehavioral symptomatology compared to published normative data (Soble et al. 2014), with at least one cognitive symptom (e.g., a score of 3 or greater on at least one of the four items on the NSI cognitive domain).

Exclusion Criteria:

* • History of TBI (any severity) within 3 months of enrollment.

  * History of moderate, severe, or penetrating TBI as defined by DOD/VA guidelines during their lifetime
  * Current substance use disorder based on patient self-report.
  * History of a neurological disease other than mild TBI such as multiple sclerosis, cerebral vascular accident, brain tumor, neurodegenerative disease, or neuro-motor disorder.
  * Current, active suicidal or homicidal ideation.
  * Impaired decision-making capacity.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 162 (Estimated)
Dates: Start 2021-02-01 (Estimated); Primary Completion 2024-09-30 (Estimated); Study Completion 2024-09-30 (Estimated)

PRIMARY OUTCOMES:
Change in cognitive impairment | 4 MONTHS
  Cognitive impairment will be measured using the Global Deficit Score (GDS) which allows for the detection of subtle and varied degree of impairment from multiple measures.

SECONDARY OUTCOMES:
Change in healthcare utilization | 4.5 MONTHS
  Healthcare utilization post-treatment, as measured by the number of medical appointments to rehabilitation specialists.
Change in level of occupational performance | 4.5 MONTHS
  Ratings of occupational performance by a direct supervisor using a modified Checklist of Military Activities of Daily Living (M-ADL).

CONTACTS AND LOCATIONS:
Locations (1):
- Naval Hospital Camp Pendleton, Oceanside, California, United States

IPD SHARING:
Plan to Share IPD: No